CLINICAL TRIAL: NCT00189826
Title: A Multicentre, Randomised, Double Blind, Two Arm Parallel Group Study to Evaluate and Compare the Efficacy and Safety of Modified Release Tacrolimus FK506E (MR4) Versus Tacrolimus FK506 in Combination With Steroids in Patients Undergoing Primary Liver Transplantation
Brief Title: A Study to Evaluate the Safety and Efficacy of FK506E (MR4) in Patients Undergoing Primary Liver Transplantation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FG-506E-11-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Liver Transplantation
Keywords: Tacrolimus; Liver transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tacrolimus
- 2 (Experimental)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — immunosuppression
  Other Names: FK506E, MR4

SUMMARY:
To evaluate and to compare efficacy and safety of a dual regimen with oral modified release tacrolimus FK506E (MR4) / steroids versus a dual regimen with oral tacrolimus FK506 / steroids in patients undergoing primary liver transplantation. It shall be demonstrated that FK506E (MR4) is non-inferior to FK506 with regards to the primary endpoint.

DETAILED DESCRIPTION:
A multicentre, 1:1 randomised, double blind, double dummy, two arm parallel group phase III study comparing a dual modified release FK506E (MR4) / steroid regimen with a standard tacrolimus FK506 / steroid regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a primary, split liver or a whole liver graft from a cadaveric donor with compatible ABO blood type.

Exclusion Criteria:

* Patients receiving a multi-organ transplant or having previously received an organ transplant (including liver re-transplantation).
* Patients with severe diarrhoea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus.
* Patients with serum creatinine > 200 µmol/l..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2004-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Incidence of and time to biopsy-proven acute rejections | 12 months

SECONDARY OUTCOMES:
Incidence of acute rejections | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: J. Langrehr, Principal Investigator — Charite Campus Virchow Klinikum
Locations (49):
- Australia (2):
  - Heidelberg
  - Sydney
- Belgium (2):
  - Ghent
  - Liège
- Brazil (4):
  - Bel Horizonte
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (5):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Prague, Czechia
- Helsinki, Finland
- France (8):
  - Clichy
  - Créteil
  - Lyon
  - Montpellier
  - Rennes
  - Strasbourg
  - Toulouse
  - Villejuif
- Germany (4):
  - Berlin
  - Hamburg
  - Heidelberg
  - Regensburg
- Dublin, Ireland
- Italy (6):
  - Bergamo
  - Bologna
  - Genova
  - Modena
  - Palermo
  - Udine
- Oslo, Norway
- Warsaw, Poland
- Spain (6):
  - Barakaldo
  - Barcelona
  - Córdoba
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (2):
  - Gothenburg
  - Stockholm
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (3):
  - Leeds
  - London
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Ericzon BG, Varo E, Trunecka P, Fischer L, Colledan M, Gridelli B, Valdivieso A, O'Grady J, Dickinson J, Undre N. Pharmacokinetics of prolonged-release tacrolimus versus immediate-release tacrolimus in de novo liver transplantation: A randomized phase III substudy. Clin Transplant. 2017 Jun;31(6). doi: 10.1111/ctr.12958. Epub 2017 Apr 27. PMID 28295581